CLINICAL TRIAL: NCT04549415
Title: The Effect of Metformin on Clinical Course of Ischemic Etiology Chronic Heart Failure in Patients With Prediabetes: the Open-label Randomized Clinical Trial
Brief Title: The Influence of Metformin on Chronic Heart Failure Clinical Course in Patients With Prediabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government)
Responsible Party: Principal Investigator, Bermet Kurmanbekova, Principal investigator, researcher in chronic heart failure department, National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NoruzbaevaCHF
Record Dates: First submitted 2020-09-03; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Chronic Heart Failure; Coronary Artery Disease; PreDiabetes
Keywords: metformin; chronic heart failure; prediabetes; insulin resistance; clinical course
MeSH Terms: conditions — Coronary Artery Disease; Prediabetic State; Insulin Resistance; Disease Progression | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- metformin (Active Comparator): Metformin, 1000 mg b.i.d, 12 months
  Interventions: Drug: Metformin Hydrochloride
- lifestyle modification (Active Comparator): Lifestyle modification Standard Principles
  Interventions: Other: lifestyle modification

INTERVENTIONS:
Drug: Metformin Hydrochloride — patients were divided into 2 groups: 1st group was on lifestyle modification (LSM), 2nd group on regimen "LSM+ metformin (1000 g b.i.d)" during 12 months
  Arms: metformin
Other: lifestyle modification — Lifestyle modification Standard Principles
  Arms: lifestyle modification

SUMMARY:
It is well known fact, that prediabetes is a predictor of high cardiovascular mortality, increasing the risk of developing such adverse cardiovascular events as myocardial infarction, stroke and sudden cardiac death. The key pathogenetic link in development of carbohydrates metabolism disorders (CMD) is insulin resistance (IR), which is one of the crucial mechanisms for the development and progression of chronic heart failure (CHF). IR disrupts the functioning of the myocardium due to endothelial dysfunction, inflammation, oxidative stress, remodeling and impaired myocardial metabolism. In condition of a combination of CMD and CHF the reverse development of hyperglycemia is also difficult due to hyperactivation of neurohormonal systems - renin-angiotensin-aldosterone system, in particular.

So, drug therapy should neutralize the undesirable metabolic effects of hyperglycemia on the course of CHF, as well as prevent the development of micro- and macrovascular complications.

The study will investigate the ability of metformin to impact on clinical and laboratory (neurohormonal, lipid profiles, renal function) parameters of ischemic etiology heart failure patients with prediabetes, as well as their quality of life and prognosis (incidence of adverse cardiovascular events). These tests will be assessed at the beginning and repeated after one year. At the end of the study we will investigate the difference between lifestyle modification effect and metformin treatment.

The study is funded by Ministry of Education and Science of Kyrgyz Republic.

DETAILED DESCRIPTION:
This is a single centre trial designed to investigate the benefit, if any, of 12-month metformin 2000 mg/day treatment on clinical course of chronic heart failure in 78 patients with coronary artery disease and impaired glucose tolerance.

Participants will be seen in three occasions: screening, baseline randomization, 6 month, final 12 month, during which clinical and laboratory indicators will be assessed. There will also be three telephone visits at: month 1, month 3, month 9.

At a screening visit an initial history will be performed during following informed consent. Participants will undergo a laboratory, clinical and instrumental screening in Chronic Heart Failure department of National Centre of cardiology and Internal Medicine named after academician M.Mirrakhimov. Among with anthropologic and clinical data, prior to metformin administration, blood samples were evaluated.

Participants who meet all inclusion criteria will return for the randomization during hospitalization to either Metformin or Lifestyle modification alone.

After 6 months of observation safety indicators will be evaluated, as well as fasting and postprandial glucose, creatinine, ECG.

In the active arm, therapy will be metformin in an initial dose of 1000 mg/day (metformin 500 mg х2/day). Participants will continue on Metformin 500 mg x2/day for 2 weeks, following safety blood checks this dose will be increased to 2000 mg/day. If the higher dose cannot be tolerated it will be reduced to 1000 mg/day (or stopped if not tolerated).

The target dose of Metformin at 2000 mg/day was chosen based on previous study of metformin in nondiabetic heart failure patients with IR

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over (not older 65 y.o)
* Participant willing and able to give informed consent
* Documented Coronary artery disease (CAD): either angio-graphically documented CAD or a previous history of myocardial infarction/angina.
* Verified heart failure functional class III (Nt-proBNP levels, 6-min walking test)
* Fasting insulin resistance ≥ 2.5 (HOMA-IR)
* Receiving basic therapy for CAD and chronic heart failure (CHF)
* Able (in the investigators opinion) and willing to comply with all study requirements

Exclusion Criteria:

* Cognitive impairments
* Type 1 or 2 Diabetes mellitus, antihyperglycemic therapy in anamnesis
* Unstable course of CAD
* Acute heart failure or CHF decompensation
* Malignancy (receiving active treatment) or other life threatening disease
* Renal dysfunction (stage 3B or worse)
* Thyroid dysfunction
* Pregnancy/lactating females
* Any other reason considered inappropriate by a study physician
* Participants who have participated in any other clinical trial within the previous 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 12 months
  Safety and efficacy of Metformin will be determined by monitoring changes from randomization till the end of the study or so long the patient remains in the study , whichever is earlier
Number of participants with newly diagnosed diabetes mellitus | 12 months
  Carbohydrate metabolism indicators will be determined by monitoring changes in fasting, postprandial glycemia and glycated hemoglobin

SECONDARY OUTCOMES:
Chronic heart failure patients Quality of Life | 12 months
  Minnesota Living with Heart Failure Questionnaire will be evaluated at baseline and at 12 months
6-minute walking test results | 12 months
  The test is based on measuring the walking distance with turns along a long corridor (≥30 m) at the patient's own pace. Results will be evaluated at baseline and at 12 months
Insulin resistance by HOMA-IR | 12 months
  Improvement in insulin (insulin resistance by HOMA-IR) when treated with metformin compared to lifestyle modification in patients with ischemic etiology CHF and prediabetes using ELISA
Aldosterone levels | 12 months
  Improvement in aldosterone levels when treated with metformin compared to lifestyle modification in patients with ischemic etiology CHF and prediabetes using ELISA
Nt-proBNP levels | 12 months
  Improvement in Nt-proBNP levels when treated with metformin compared to lifestyle modification in patients with ischemic etiology CHF and prediabetes using ELISA
Renal function markers | 12 months
  Creatinine levels with estimated glomerular filtration rate and daily proteinuria at a baseline and at 12 months to assess safety and influence of metformin
Lipid profile markers | 12 months
  Improvement in lipid profile indicators (total cholesterol, high- and low-density lipoprotein cholesterol, triglycerides) when treated with metformin compared to lifestyle modification

CONTACTS AND LOCATIONS:
Overall Officials: Akbay Sarybaev, Study Director — National Centre of Cardiology and Internal Medicine
Locations (1):
- National Centre of Cardiology and Internal Medicine named after academician M.Mirrakhimov, Bishkek, Kyrgyzstan